CLINICAL TRIAL: NCT00326885
Title: A Single-Arm, Open-Label, Phase II Study to Assess the Safety and Efficacy of the Trifunctional Antibody Catumaxomab (Anti-EpCAM x Anti-CD3) Administered Intraperitoneally in Ovarian Cancer Patients With Recurrent Symptomatic Malignant Ascites
Brief Title: Study of the Trifunctional Antibody Catumaxomab to Treat Recurrent Symptomatic Malignant Ascites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Collaborators: Fresenius Biotech North America (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-REM-AC-02-US
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Malignant Ascites
Keywords: Ascites; Epithelial Cancer; Epithelial Carcinoma; Epithelial Ovarian Cancer; Epithelial Ovarian Carcinoma; Fallopian Tube Cancer; Fallopian Tube Carcinoma; Malignant Ascites; Ovarian Cancer; Ovarian Carcinoma; Ovarian Epithelial Cancer; Ovarian Epithelial Carcinoma; Peritoneal Cancer; Peritoneal Carcinoma; Recurrent Ascites; Recurrent Malignant Ascites; Recurrent Symptomatic Malignant Ascites; Symptomatic Malignant Ascites; Symptomatic Ascites; Neoplasms, Glandular and Epithelial; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms
MeSH Terms: conditions — Ascites; Carcinoma; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms; Neoplasms, Glandular and Epithelial; Peritoneal Neoplasms | interventions — catumaxomab

ARMS (1):
- Catumaxomab (Experimental)
  Interventions: Drug: catumaxomab

INTERVENTIONS:
Drug: catumaxomab — Catumaxomab is administered intraperitoneally via an indwelling catheter (or port) as a 3-hour infusion 4 times (Days 0, 3, 7, and 10) in ascending doses (10 mcg, 20 mcg, 50 mcg, and 150 mcg, respectively).

SUMMARY:
The purpose of this study is to determine whether the investigational drug catumaxomab is a safe and effective treatment for recurrent symptomatic malignant ascites.

DETAILED DESCRIPTION:
A multi-center, phase II study of catumaxomab in ovarian cancer patients with recurrent symptomatic malignant ascites requiring therapeutic paracentesis. Each eligible patient will receive four ascending doses of catumaxomab, administered intraperitoneally via an indwelling catheter. Catumaxomab will be administered as a 3-hour constant rate infusion with a dosing interval of 3-4 days. Each patient will participate in this study for up to 7 months (includes the baseline therapeutic paracentesis and screening period, 11 to 21 days treatment period, and up to 180 days/6 months follow-up), with monthly post-study follow-up for the lifetime of the patient.

Catumaxomab is a trifunctional antibody targeting EpCAM on tumor cells and CD3 on T cells. Trifunctional antibodies represent a new concept for targeted anticancer therapy. This new antibody class has the capability to redirect T cells and accessory cells (e.g. macrophages, dendritic cells (DCs) and natural killer (NK) cells) to the tumor site. According to preclinical data, trifunctional antibodies activate these different immune effector cells, which can trigger a complex anti-tumor immune response.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Histologically confirmed diagnosis of epithelial ovarian cancer, peritoneal cancer, or fallopian tube cancer; any stage at diagnosis [International Federation of Gynecology and Obstetrics (FIGO) Stages I through IV].
* Progression on or ≤ 12 months after primary platinum-based systemic or intraperitoneal (IP) chemotherapy OR relapse following reinduction ≥ 12 months after primary chemotherapy.
* Have refused, failed, or have been deemed not suitable candidates for gemcitabine or liposomal doxorubicin.
* Recurrent symptomatic malignant ascites requiring therapeutic paracentesis
* At least 1 therapeutic paracentesis within 4 weeks prior to baseline paracentesis
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy ≥ 16 weeks
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN, and total bilirubin ≤ 1.5 x ULN
* Absolute neutrophil count (ANC) ≥ 1,500/mm3 and platelet count ≥ 75,000/mm3
* Negative serum pregnancy test result at screening in women of childbearing potential (applies to patients without documented menopause or sterility).
* Willingness of patients of childbearing potential to use an effective contraceptive method (i.e., oral contraceptive, cervical cap, diaphragm with spermicide, condom with spermicide, or intrauterine device) during the study and for at least 6 months after the last infusion.

Exclusion Criteria:

* Acute or chronic systemic infection
* Exposure to investigational drugs, chemotherapy or radiotherapy 21 days prior to the first dose of catumaxomab
* Major surgery 2 weeks prior to first dose
* Previous treatment with mouse or rat antibodies
* Known or suspected hypersensitivity to catumaxomab or other monoclonal antibodies
* Body mass index (BMI) < 19 (body weight after paracentesis to be used for calculation of BMI)
* Serum albumin level < 2.0 g/dL
* Reduced nutritional status requiring predominantly parenteral nutrition (> 50% of energy intake). Permanent naso-gastric (NG) feeding tube.
* Ileus in a location that precludes paracentesis
* Extensive liver metastases (> 70% organ volume comprises malignancy)
* Documented brain metastases
* History of myocardial infarction, congestive heart failure or relevant cardiac arrhythmia 3 months prior to the first dose of catumaxomab
* Portal vein obstruction or portal vein thrombosis diagnosed by computed tomography (CT) scan at screening
* Persistent massive pleural effusion or inadequate respiratory function of any other etiology (except if related to ascites symptoms) in the opinion of the investigator
* Any other condition which, according to the investigator, results in an undue risk to the patient by participating in the study
* Prior exposure to catumaxomab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Berek, MD MMSc, Study Chair — Stanford University Hospital and Clinics, Department of Obstetrics and Gynecology
Locations (18):
- United States (18):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of San Diego, La Jolla, California
  - Stanford University Hospital and Clinics, Stanford, California
  - University of Miami, Miami, Florida
  - Florida Hospital Cancer Center, Orlando, Florida
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Louisville Cancer Center, Louisville, Kentucky
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Dartmouth-Hitchock Medical Center, Lebanon, New Hampshire
  - Columbia University Cancer center, New York, New York
  - Wake-Forest University, Winston-Salem, North Carolina
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Magee Women's Hospital, University of Pittsburgh, Pittsburgh, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Background] Heiss MM, Strohlein MA, Jager M, Kimmig R, Burges A, Schoberth A, Jauch KW, Schildberg FW, Lindhofer H. Immunotherapy of malignant ascites with trifunctional antibodies. Int J Cancer. 2005 Nov 10;117(3):435-43. doi: 10.1002/ijc.21165. PMID 15906359
- [Background] Ruf P, Lindhofer H. Induction of a long-lasting antitumor immunity by a trifunctional bispecific antibody. Blood. 2001 Oct 15;98(8):2526-34. doi: 10.1182/blood.v98.8.2526. PMID 11588051
- [Background] Riesenberg R, Buchner A, Pohla H, Lindhofer H. Lysis of prostate carcinoma cells by trifunctional bispecific antibodies (alpha EpCAM x alpha CD3). J Histochem Cytochem. 2001 Jul;49(7):911-7. doi: 10.1177/002215540104900711. PMID 11410615
- [Background] Zeidler R, Mysliwietz J, Csanady M, Walz A, Ziegler I, Schmitt B, Wollenberg B, Lindhofer H. The Fc-region of a new class of intact bispecific antibody mediates activation of accessory cells and NK cells and induces direct phagocytosis of tumour cells. Br J Cancer. 2000 Jul;83(2):261-6. doi: 10.1054/bjoc.2000.1237. PMID 10901380
- [Background] Zeidler R, Reisbach G, Wollenberg B, Lang S, Chaubal S, Schmitt B, Lindhofer H. Simultaneous activation of T cells and accessory cells by a new class of intact bispecific antibody results in efficient tumor cell killing. J Immunol. 1999 Aug 1;163(3):1246-52. PMID 10415020
- [Background] Heiss MM, Murawa P, Koralewski P, Kutarska E, Kolesnik OO, Ivanchenko VV, Dudnichenko AS, Aleknaviciene B, Razbadauskas A, Gore M, Ganea-Motan E, Ciuleanu T, Wimberger P, Schmittel A, Schmalfeldt B, Burges A, Bokemeyer C, Lindhofer H, Lahr A, Parsons SL. The trifunctional antibody catumaxomab for the treatment of malignant ascites due to epithelial cancer: Results of a prospective randomized phase II/III trial. Int J Cancer. 2010 Nov 1;127(9):2209-21. doi: 10.1002/ijc.25423. PMID 20473913
- [Background] Ruf P, Kluge M, Jager M, Burges A, Volovat C, Heiss MM, Hess J, Wimberger P, Brandt B, Lindhofer H. Pharmacokinetics, immunogenicity and bioactivity of the therapeutic antibody catumaxomab intraperitoneally administered to cancer patients. Br J Clin Pharmacol. 2010 Jun;69(6):617-25. doi: 10.1111/j.1365-2125.2010.03635.x. PMID 20565453
- [Derived] Berek JS, Edwards RP, Parker LP, DeMars LR, Herzog TJ, Lentz SS, Morris RT, Akerley WL, Holloway RW, Method MW, Plaxe SC, Walker JL, Friccius-Quecke H, Krasner CN. Catumaxomab for the treatment of malignant ascites in patients with chemotherapy-refractory ovarian cancer: a phase II study. Int J Gynecol Cancer. 2014 Nov;24(9):1583-9. doi: 10.1097/IGC.0000000000000286. PMID 25254563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 patients were recruited and 32 patients were treated and evaluable. For analyses, there were 32 patients in the Full Analysis Set (FAS), 14 patients in the Per-Protocol (PP) population, and 32 patients in the Safety population.
Pre-assignment Details: Eligible patients must have undergone at least 1 therapeutic paracentesis (the most recent paracentesis) within 4 weeks prior to the baseline paracentesis.
Groups:
- Catumaxomab: Each eligible patient will receive four ascending doses of catumaxomab, administered intraperitoneally via an indwelling catheter. Catumaxomab will be administered as a 3-hour constant rate infusion with a dosing interval of 4 days (10 μg, 20 μg, 50 μg, and 150 μg, respectively)
Period: Overall Study
Arm/Group | Catumaxomab
Started | 32
Completed | 25
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Hospice withdrew consent | 2

BASELINE CHARACTERISTICS:
Arm/Group | Catumaxomab
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Achieved at Least a 4-fold Increase of Puncture/Paracentesis-free Interval Following Catumaxomab Relative to Their Pre-treatment Interval.
Description: The parameter to be estimated is the proportion of patients who achieve at least a 4-fold increase in their puncture/paracentesis-free interval. The pretreatment interval is defined as the length of time between the patient's most recent paracentesis (baseline) and the subsequent paracentesis necessitated by her increasing ascites-related symptoms. The post-treatment interval is defined as the time between the last dose of catumaxomab plus 1 day to the time of recurrence of ascites requiring therapeutic paracentesis or death, whichever occurred sooner.
Time Frame: 6 months
Measure: Number; unit: proportion of patients
Arm/Group | Catumaxomab
Number analyzed (Participants) | 31
proportion of patients | 0.226

2. Secondary Outcome: Puncture/Paracentesis-free Survival (PuFS)
Description: Puncture/Paracentesis-free Survival (PuFS), Defined as the Number of Days Between the Date of Last Dose and the Date of Documented End of Study (EoS) Paracentesis or Death, Whichever Occurred First
Time Frame: ≥6 months
Population: Full analysis set (FAS) Per protocol (PP)
Measure: Median (Full Range); unit: weeks
Arm/Group | Catumaxomab
Number analyzed (Participants) | 32
weeks | 4.2 [2.1 to 7.6]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the interval from the date of first dose to the date of death.
Time Frame: ≥ 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Catumaxomab
Number analyzed (Participants) | 32
months | 3.6 [2.2 to 4.6]

4. Secondary Outcome: Ascites Signs and Symptoms
Description: Patient-reported ascites symptoms were to be assessed using the patient questionnaire, Functional Assessment of Chronic Illness Therapy - Ascites Index (FACIT-AI). At 6 months following catumaxomab administration, the patient was requested to assess the severity of the following parameters during the past week using a 5-point scale with scores from "0 = not at all" to "4 = very much": anorexia, insomnia, decreased mobility, dyspnea, nausea, vomiting, abdominal pain, abdominal distention, fatigue, early satiety, urinary frequency, constipation, and emotional distress. For the parameters anorexia, insomnia, and decreased mobility, high scores mean good response, for the other parameters low scores mean good response.
Time Frame: 6 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Catumaxomab
Number analyzed (Participants) | 4
units on a scale
  I have good appetite | 1.5 [1 to 2]
  I am sleeping well | 1.0 [1 to 2]
  I am able to get around by myself | 1.0 [0 to 3]
  I have been short of breath | 1.0 [1 to 1]
  I have nausea | 0.5 [0 to 2]
  I have been vomiting | 0.5 [0 to 1]
  I have pain in my stomach area | 1.0 [1 to 1]
  I have swelling in my stomach area | 1.0 [0 to 2]
  I have lack of energy | 2.0 [1 to 3]
  When I eat, I seem to get full quickly | 2.0 [2 to 3]
  I urinate more frequently | 0.0 [0.0 to 2.0]
  I am bothered by constipation | 1.0 [0 to 1]
  I have been emotionally distressed | 0 [0 to 0]

5. Secondary Outcome: Ascites Volume
Description: Ascites volume measurement were to be performed at screening (= prior to baseline), at baseline (= before start of therapy with catumaxomab) and during the 6-month follow-up period when the patient had recurrence of symptomatic ascites requiring therapeutic paracentesis. At each paracentesis, drainage to dryness was to be achieved and the exact volume was to be measured and documented.
Time Frame: 6 months
Measure: Median (Full Range); unit: mL
Arm/Group | Catumaxomab
Number analyzed (Participants) | 32
mL
  prior to baseline (at screening) | 2800 [50 to 8675]
  baseline (start of therapy) | 2050 [60 to 5500]
  at puncture visit/ end of study (day 180) | 1500 [0 to 3100]

6. Primary Outcome: Increase of Paracentesis/Puncture-free Interval (Ratio)
Description: The parameter to be tested is the ratio of the post-treatment puncture/paracentesis-free interval divided by the pre-treatment puncture/paracentesis-free interval. The pre-treatment interval is defined as the length of time between the patient's most recent paracentesis (baseline) and the subsequent paracentesis necessitated by her increasing ascites-related symptoms. The post-treatment interval is defined as the time between the last dose of catumaxomab plus 1 day to the time of recurrence of ascites requiring therapeutic paracentesis or death, whichever occurred sooner.
Time Frame: 180 days
Measure: Median (Full Range); unit: fold
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 31
fold | 2 [0.15 to 60]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Catumaxomab
Serious Adverse Events (participants affected / at risk) | 24/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catumaxomab (N=32)
Vomiting (Gastrointestinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 5 (7)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Extravasation (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Device leakage (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (2)
Sepsis syndrome (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catumaxomab (N=32)
Anaemia (Blood and lymphatic system disorders) | 10 (10)
Tachycardia (Cardiac disorders) | 5 (6)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Diplopia (Eye disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 24 (39)
Vomiting (Gastrointestinal disorders) | 24 (37)
Abdominal pain (Gastrointestinal disorders) | 16 (19)
Constipation (Gastrointestinal disorders) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 9 (11)
Abdominal distension (Gastrointestinal disorders) | 5 (6)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 19 (21)
Pyrexia (General disorders) | 19 (34)
Chills (General disorders) | 14 (22)
Oedema peripheral (General disorders) | 9 (12)
Asthenia (General disorders) | 6 (6)
Catheter site pain (General disorders) | 5 (6)
Oedema (General disorders) | 4 (5)
Performance status decreased (General disorders) | 3 (3)
Catheter site erythema (General disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Device leakage (General disorders) | 2 (2)
Extravasation (General disorders) | 2 (2)
Candidiasis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 4 (4)
Haemoglobin decreased (Investigations) | 4 (5)
Weight decreased (Investigations) | 4 (4)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
C-reactive protein increased (Investigations) | 3 (3)
Haematocrit decreased (Investigations) | 3 (4)
Protein total decreased (Investigations) | 3 (3)
Blood albumin decreased (Investigations) | 2 (2)
Blood chloride decreased (Investigations) | 2 (2)
Blood magnesium decreased (Investigations) | 2 (2)
Coagulation time prolonged (Investigations) | 2 (2)
Oxygen saturation decreased (Investigations) | 2 (2)
Urine output decreased (Investigations) | 2 (2)
White blood cell count increased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 11 (13)
Dehydration (Metabolism and nutrition disorders) | 10 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Polydipsia (Metabolism and nutrition disorders) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 3 (6)
Tremor (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 5 (5)
Confusional state (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 2 (3)
Renal failure (Renal and urinary disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (5)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Site may publish the results of the Study after such cooperative publication, or 1 year after Sponsor's final evaluation of all the Study data from all sites, whichever occurs first. Prior to any submission for publication, presentation, or communication of results or information arising from the Study, Investigator shall provide Fresenius Biotech at least 90 days for review and comment upon the manuscript or other material for such publication or presentation.